CLINICAL TRIAL: NCT03767764
Title: Yliver as a Test to Early Diagnose Hepatocellular Carcinoma
Brief Title: Yliver as a Test to Early Diagnose HCC
Acronym: YliverDIAG
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Juan Francisco Delgado de la Poza, Senior Immunologist, Corporacion Parc Tauli
Other Study IDs: CIR2017/024
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Tumor associated antigen; Early diagnosis; Autoantibodies; Alpha fetoprotein
MeSH Terms: conditions — Carcinoma, Hepatocellular; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HCC: Patients with diagnosis of Hepatocellular carcinoma
  Interventions: Diagnostic Test: Test Yliver
- Cirrhosis: Patients with the diagnosis of cirrhosis who is following a screening program for diagnosis of HCC
  Interventions: Diagnostic Test: Test Yliver
- Chronic liver diseases: Patients with the diagnosis of Chronic liver diseases without cirrhosis
  Interventions: Diagnostic Test: Test Yliver
- Control: Normal human serum from donors without liver disease
  Interventions: Diagnostic Test: Test Yliver

INTERVENTIONS:
Diagnostic Test: Test Yliver — Test Yliver is used to detect autoantibodies against alpha fetoprotein in serum by an ELISA technique

SUMMARY:
Liver cancer (HCC) is the second cause of death related to cancer worldwide, with about 750,000 deaths from this cause in 2012. Although the early diagnosis of liver cancer increases the available treatment options, the methods currently used for screening are not sufficiently sensitive for this purpose.

The investigators provide a high-performance and highly reliable in vitro platform that allows the identification and quantification of autoantibodies in serum for use as biomarkers of liver cancer, using an ELISA test (Yliver).

The aim of the study is to demonstrate whether the Yliver test can be used as a biomarker for the early diagnosis of hepatocellular carcinoma with a collection of samples from 58 patients diagnosed with HCC, 42 cirrhosis, 40 normal controls and the inclusion of 25-50 patients with chronic liver disease without cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

EASL Clinical Practice Guidelines & Practice Guidance by the American Association for the Study of Liver Diseases for diagnosis of HCC, liver cirrhosis, chronic hepatitis without cirrhosis

Exclusion Criteria:

* Age under 18 years
* Very advanced disease (patient in a terminal state that is not indicated analytical determinations).
* Hepatic encephalopathy that prevents the correct understanding of informed consent.
* Refusal to carry out the determination or to sign the informed consent.
* Patients affected by another neoplastic disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HCC: patients with HCC diagnosis Cirrhosis: patients with liver cirrhosis diagnosis Chronic liver disease: patients with chronic liver diasease without cirrhosis Control: normal human serum from donors without liver disease
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Yliver | October 2018-February 2019
  Titer of autoantibodies against alpha fetoprotein applying Taby Technology

SECONDARY OUTCOMES:
AFP | October 2018-February 2019
  Levels of alpha fetoprotein in serum
Ultrasound | October 2018-February 2019
  Results of the ultrasound examination
AAb AFP | October 2018-February 2019
  Titer of autoantibodies against alpha fetoprotein with standard protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Corporacion Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No